CLINICAL TRIAL: NCT00874627
Title: Sublingual Milk Immunotherapy in Children With IgE-mediated Cow Milk Protein Allergy
Brief Title: Sublingual Milk Immunotherapy in Children
Acronym: Lactaide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ESPCI Paris (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K070602
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Cow Milk Allergy
Keywords: children > 5 years old; IgE-mediated; cow milk allergy; IgE-mediated cow milk allergy persisting after 5 years
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Administration of Milk
  Interventions: Other: Milk
- Placebo (Placebo Comparator): meals without milk
  Interventions: Other: Milk

INTERVENTIONS:
Other: Milk — sublingual administration of milk
  Other Names: sublingual administration of milk
  Arms: Experimental
Other: Milk — placebo
  Other Names: placebo
  Arms: Placebo

SUMMARY:
Sublingual immunotherapy is developing in the treatment of aeroallergens allergy. The hypothesis is that such process may be applied to food allergy, more precisely to milk. A previous series of 8 patients indicates the likely effectiveness of this technique (Allergy, 2006).

DETAILED DESCRIPTION:
National study of current practice, multicentric, randomized, open All oral provocation tests will be randomized, double blind Study treatment. For oral provocation test, placebo with NeocatePasteurized half skimmed milk (available in standard outlets) from 0.1 to 0.8 mL/day Tests At M0 :1) Clinical examination 2) Biological test (blood sample 16.5 mL) : WBC, ferritin, total IgE, specific IgE, cow milk, ALPHALACTALBUMIN , casein, BETALACTOGLOBULIN and goat milk using RASTSpecific secretory IgA by ESPCI (frozen saliva)Biologic collection- Specific immunoglobulins against cow' milk, ALPHALACTALBUMIN, casein, BETALACTOGLOBULIN, quantification of IgM, sub classes of IgG and IgA by ESPCI (frozen serum).

Analysis of minor allergens by immunoblot 2 D, ESPCI (frozen serum)3) prick tests 4) 1 or 2 oral provocation test (TPO) double blind, during 2 days At M3 : clinical examination, side effects during the 3 preceding months At M6 :1) Clinical examination 2) Biological test (blood sample 16.5 mL) : WBC, ferritin, total IgE, specific IgE, cow milk, ALPHALACTALBUMIN, casein, BETALACTOGLOBULIN and goat milk using RAST Specific secretory IgA by ESPCI (frozen saliva)Biologic collection Specific immunoglobulins against cow' milk, ALPHALACTALBUMIN, casein, BETALACTOGLOBULIN, quantification of IgM, sub classes of IgG and IgA by ESPCI (frozen serum).

Analysis of minor allergens by immunoblot 2 D, ESPCI (frozen serum)3) prick tests 4) 1 or 2 oral provocation test (TPO) double blind, during 2 days At M12 :1) Clinical examination2) Biological test (blood sample 16.5 mL) : WBC, ferritin, total IgE, specific IgE, cow milk, ALPHALACTALBUMIN, casein, BETALACTOGLOBULIN and goat milk using RAST Specific secretory IgA by ESPCI (frozen saliva)Biologic collection- Specific immunoglobulins against cow' milk, ALPHALACTALBUMIN, casein, BETALACTOGLOBULIN , quantification of IgM, sub classes of IgG and IgA by ESPCI (frozen serum).

Analysis of minor allergens by immunoblot 2 D, ESPCI (frozen serum)3) prick tests 4) 1 or 2 oral provocation test (TPO) double blind, during 2 days

ELIGIBILITY:
Inclusion Criteria:

* Children, male and female
* Children > 5 years
* Children with IgE-mediated cow milk allergy, with detectable specific IgE (> 0.10 KU/l) and an immediate type reaction during oral provocation test for a cumulated dose < 100 mL of milk).
* Children and parents or tutors having given their informed consent after complete information

Exclusion Criteria:

* Children participating or having already participated to a drug trial during the 3 preceding months
* Children with immune deficiency
* Children with disabling disease, preventing from a correct practice of sublingual treatment
* Children receiving steroid therapy
* Children refusing to participateSevere food neophobia
* Reaction to placebo during the double blind oral provocation test
* Severe anaphylactic reaction with milk during the 6 preceding months

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reactive milk dose at inclusion, at 6 months and at 12 months | at inclusion, at 6 months and at 12 months

SECONDARY OUTCOMES:
Skin reaction at inclusion at 6 months and at 12 months | at inclusion at 6 months and at 12 months
Specific IgE rate at inclusion, at 6 months and at 12 months | at inclusion, at 6 months and at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Dupont, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hospital Cochin - Saint-Vincent de Paul, Paris, France